CLINICAL TRIAL: NCT00083057
Title: A Pilot Phase I Dose Escalation Study Of The EGFR Tyrosine Kinase Inhibitor Gefitinib (Iressa) Combined With Paclitaxel (Taxol) And External Beam Radiation Therapy In Patients With Advanced Squamous Cell Carcinoma Of The Head And Neck (SCCHN)
Brief Title: Gefitinib, Paclitaxel, and Radiation Therapy in Treating Patients With Advanced or Recurrent Squamous Cell Carcinoma of the Head and Neck
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 040141; 04-C-0141; CDR0000362055; NCT00080249 (obsolete NCT alias)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Gefitinib; Paclitaxel; Radiotherapy

INTERVENTIONS:
Drug: gefitinib
Drug: paclitaxel
Radiation: radiation therapy

SUMMARY:
RATIONALE: Gefitinib may stop the growth of tumor cells by blocking the enzymes necessary for their growth. Drugs used in chemotherapy, such as paclitaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Giving gefitinib and paclitaxel together with radiation therapy may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of gefitinib and paclitaxel when given together with radiation therapy in treating patients with advanced or recurrent squamous cell carcinoma (cancer) of the head and neck.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the dose-limiting toxicity, toxicity profile, and maximum tolerated dose (MTD) of gefitinib and paclitaxel administered with radiotherapy in patients with advanced or recurrent squamous cell carcinoma of the head and neck.

Secondary

* Determine the efficacy of this regimen in patients treated at the MTD.

OUTLINE: This is a pilot, dose-escalation study of gefitinib and paclitaxel.

Patients receive oral gefitinib once daily beginning on day 1 and continuing until completion of radiotherapy. Patients receive paclitaxel IV over 1 hour on days 8, 15, 22, 29, 36, and 43 and undergo radiotherapy once daily on days 8-12, 15-19, 22-26, 29-33, 36-40, 43-47, 50-54, and 57-61. Treatment continues in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of gefitinib and paclitaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A cohort of 6 additional patients receive treatment at the MTD.

Patients are followed monthly for 1 year, every 2 months for 1 year, and then every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 15-30 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell (epidermoid) carcinoma of the oral cavity, oropharynx, hypopharynx, larynx, nasopharynx, or maxillary sinus

  * Stage III or IV disease
  * Distant metastases allowed provided both of the following are true:

    * Metastases are confined to the head and neck region
    * Metastases are encompassable in a radiotherapy field with curative intent
* Locally recurrent disease after primary surgery allowed
* Meets 1 of the following criteria:

  * Unresectable disease
  * Patient prefers chemoradiotherapy over surgery
* Measurable disease
* No brain metastases and/or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* WBC ≥ 3,000/mm^3
* Hemoglobin > 10 g/dL
* Platelet count > 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3

Hepatic

* Bilirubin < 2.0 times upper limit of normal (ULN)
* AST/ALT ≤ 2.5 times ULN

Renal

* Creatinine < 1.5 times ULN OR
* Creatinine clearance ≥ 60 mL/min

Cardiovascular

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Pulmonary

* No clinically active interstitial lung disease

  * Chronic, stable, asymptomatic radiographic changes allowed

Other

* No prior allergic reaction attributed to compounds of similar chemical or biological composition to study drugs or Cremophor^® EL
* No AIDS or primary immunodeficiencies
* No other malignancy within the past 5 years except curatively treated squamous cell or basal cell skin cancer or carcinoma in situ of the cervix

  * Probability of recurrence of the prior malignancy < 5%
* No other concurrent uncontrolled illness
* No ongoing or active serious infection
* No psychiatric illness or situation that would preclude study compliance or giving informed consent
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy for cancer
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* No prior therapeutic radiotherapy to the head and neck region
* No prior radiotherapy for cancer

Surgery

* See Disease Characteristics
* At least 4 weeks since prior major surgery and recovered

Other

* No prior gefitinib or other epidermal growth factor receptor inhibitors
* More than 4 weeks since prior non-approved or investigational agents
* No concurrent administration of any of the following:

  * Phenytoin
  * Carbamazepine
  * Barbiturates
  * Rifampin
  * Hypericum perforatum (St. John's wort)
  * Oxcarbazepine
  * Rifapentine
  * Amifostine
  * Modafinil
  * Other CYP3A4 enzyme inducers
  * Other anticancer agents or investigational drugs
  * Combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2004-05; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) and maximum tolerated dose (MTD) as assessed by CTC v. 3.0

SECONDARY OUTCOMES:
Molecular targets analysis of epidermal growth factor receptor (EGFR) downstream signaling pathway as assessed by tissue biopsies and serum cytokines at baseline, days 8 and 29, and 12 weeks after completion of study treatment
Efficacy as assessed by imagining, histologically, and clinically at 3 months after completion of study treatment and annually for 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Carter Van Waes, MD, PhD, Study Chair — National Institute on Deafness and Other Communication Disorders (NIDCD); John C. Morris, MD, Principal Investigator — NCI - Metabolism Branch;MET
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Metabolism Branch;MET, Bethesda, Maryland

REFERENCES:
- [Result] Van Waes C, Allen CT, Citrin D, Gius D, Colevas AD, Harold NA, Rudy S, Nottingham L, Muir C, Chen Z, Singh AK, Dancey J, Morris JC. Molecular and clinical responses in a pilot study of gefitinib with paclitaxel and radiation in locally advanced head-and-neck cancer. Int J Radiat Oncol Biol Phys. 2010 Jun 1;77(2):447-54. doi: 10.1016/j.ijrobp.2009.05.037. Epub 2009 Oct 30. PMID 19879702
- [Result] Sharp H, Morris JC, Van Waes C, Gius D, Cooley-Zgela T, Singh AK. High incidence of oral dysesthesias on a trial of gefitinib, Paclitaxel, and concurrent external beam radiation for locally advanced head and neck cancers. Am J Clin Oncol. 2008 Dec;31(6):557-60. doi: 10.1097/COC.0b013e318172d5de. PMID 19060587
- [Result] Sharp HJ, Morris JC, Van Waes C, et al.: A high incidence of oral dysesthesias unrelated to mucositis in a pilot trial of gefitinib, paclitaxel and concurrent external beam radiation in patients with locally advanced squamous cell carcinoma of the head and neck (SCCHN). [Abstract] Int J Radiat Oncol Biol Phys 66 (3 Suppl 1): A-1101, S188-9, 2006.